CLINICAL TRIAL: NCT02326571
Title: Multimodal Monitoring in Patients With Spontaneous Intracerebral Hemorrhage
Status: Completed | Type: Observational
Sponsor: Christian Kærsmose Friberg (Other)
Responsible Party: Sponsor-Investigator, Christian Kærsmose Friberg, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-1-2014-059
Record Dates: First submitted 2014-12-12; First posted 2014-12-29 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Hemorrhage
Keywords: EEG; Cortical Spreading Depression; Cerebral Hemorrhage; miRNA; Reactivity in EEG; Multimodal monitoring
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For later miRNA analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- spontaneous intracerebral hemorrhage

SUMMARY:
Spontaneous intracerebral bleeding also known as spontaneous intracerebral hemorrhage (sICH) constitute 10-15 % of all apoplexies. The Prognosis is considerably worse than it is for the larger population of patients suffering from cerebral thrombosis. Development of brain edema seemingly contributes to the disadvantageous prognosis. However, the mechanisms behind is only understood fragmentarily.

By using multimodal neuro monitoring, the investigators seek to investigate electrophysiological and metabolic processes, which seem to accompany the formation of edema and clinical deterioration in patients suffering from sICH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: spontaneous intracerebral hemorrhage verified by CT
* Clinical indication for craniotomy or craniectomy
* Admitted to the hospital within 24 hours from assumed ictus
* Age over 18 years

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for neuro surgery admitted to Rigshospitalet, Copenhagen with spontaneous intracerebral hemorrhage verified by CT.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Secondary brain injury | 10 days
  Assessed by GCS, CAM-ICU, mRS, Imaging, EEG background activity.

CONTACTS AND LOCATIONS:
Overall Officials: Christian K Friberg, MD, Principal Investigator
Locations (1):
- Rigshospitalet, NICU, Copenhagen, Denmark